CLINICAL TRIAL: NCT02482467
Title: Prognosis and Long Term Pubertal Outcome of Girls Previously Diagnosed With a Prenatal Ovarian Cyst
Acronym: KYSTOV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No difference between groups after analysis
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9434; 2014-A01025-42 (Registry Identifier: ID RCB)
Record Dates: First submitted 2015-06-15; First posted 2015-06-26 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cyst
Keywords: ovarian cyst; prenatal diagnosis; puberty
MeSH Terms: conditions — Ovarian Cysts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cases (Other): Prenatal diagnosis of ovarian cyst
  Interventions: Other: Hormonal analysis, pelvic US
- controls (Other): No prenatal diagnosis of cyst
  Interventions: Other: Hormonal analysis, pelvic US

INTERVENTIONS:
Other: Hormonal analysis, pelvic US

SUMMARY:
Puberty and long-term ovarian function of patients with a ovarian prenatal cyst has not described to date.

DETAILED DESCRIPTION:
The prenatal diagnosis of ovarian cysts is a common disease with an estimated incidence of 1 case per 2500 births. This pathology is the first diagnosis of abdominal cystic picture on the female fetus in the third trimester of pregnancy.Various complications of ovarian cysts have been described, such as ovarian torsion, breaking the cyst, hemorrhage intra cystic and compression of adjacent viscera. A conservative attitude for uncomplicated cysts is proposed in the literature but surgical care and / or puncture can be made to prevent the occurrence of complications and thus to protect ovarian tissue.However, no data on puberty and long-term ovarian prognosis in this disease is published in the literature. Without this information, no support for the recommendation of a prenatal ovarian cyst can be established formally.

ELIGIBILITY:
Inclusion Criteria:

* Collection of the written consent by the patients or the parents
* Membership in a health insurance scheme
* Group 1 : girl with prenatal ovarian cyst group 2: girl without prenatal ovarian cyst

Exclusion Criteria:

* Refusal of participation of the patient or one of the two parents
* Deprived of freedom
* Pregnancy and current feeding
* Prenatal, neonatal or infantile history of ovarian pathology (Group 2)
* Genital congenital deformation or malformation syndrome gives a complex (group 2)
* Endocrine pathology except the juvenile disorders (group 2)

Ages: 6 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Age of puberty | 1 day
  Clinical data and clinical history

SECONDARY OUTCOMES:
Follicular reserve | 1 day
  Serum level of Anti-Mullerian Hormone and ovarian volume at ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas KALFA, MD, PhD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Hôpital Lapeyronie, Montpellier, France